CLINICAL TRIAL: NCT07354971
Title: The Immuno-FIT Observational Study: A Phase II Window Observational Study Investigating the Effects of Immunotherapy on Cardiopulmonary Fitness, Quality of Life, and Treatment Outcomes in Patients With Advanced Cancer
Brief Title: IMMUNO-FIT Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM CAN1905; 25/SC/0293 (Other: REC); 356874 (Other: IRAS)
Record Dates: First submitted 2025-11-24; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; Immunotherapy; Physical Fitness; Quality of Life; Drug-Related Side Effects and Adverse Reactions
Keywords: Immunotherapy; Immune Checkpoint Inhibitors; Physical Fitness; Cardiopulmonary Exercise Testing; Quality of Life; Immune-Related Adverse Events; Cancer; Exercise Physiology; Tumour Microenvironment; PD-1; PD-L1; CTLA-4; Observational Study
MeSH Terms: conditions — Neoplasms; Drug-Related Side Effects and Adverse Reactions; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (plasma, serum, PBMCs) and tumour tissue (from optional research biopsies in mechanistic sub-study, n≤10) will be retained for 10 years in an HTA-licensed biobank for potential future research with appropriate ethical approval.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Study - No Study Intervention — This is an observational study with no study-assigned interventions. All participants receive standard-of-care immunotherapy as prescribed by their treating oncologist. Immunotherapy may include anti-PD-1, anti-PD-L1, anti-CTLA-4 agents, or approved combination regimens. All doses, schedules, treatment modifications, delays, and discontinuations follow routine clinical practice and manufacturer guidance. Treatment decisions are made independently of the study. The study observes and records treatment administration, effects on fitness and quality of life, adverse events, and clinical outcomes without influencing clinical care.
  Other Names: Standard of Care Immunotherapy

SUMMARY:
This observational study will investigate how immunotherapy affects physical fitness, quality of life, and treatment tolerance in adults with solid cancers. Immunotherapy can cause a range of side effects that impact daily functioning and may lead to treatment delays or early discontinuation. Physical fitness may influence how well patients cope with treatment, yet little is known about how fitness changes during immunotherapy or whether baseline fitness is linked to outcomes.

Participants will complete fitness testing using cardiopulmonary exercise testing (CPET) and quality-of-life questionnaires before starting immunotherapy and again 12 weeks later. Blood samples will also be taken, and long-term outcomes including survival, disease progression, and quality of life will be followed for up to 24 months. All cancer treatment will remain standard of care.

A small number of participants will be invited to take part in an optional research biopsy at week 12 to explore how physical fitness relates to changes in the tumour's immune environment.

The study will help researchers understand natural changes in fitness during immunotherapy, identify whether baseline fitness is associated with treatment tolerance or outcomes, and generate information needed to design future trials testing exercise-based interventions during immunotherapy.

DETAILED DESCRIPTION:
Physical fitness is a strong prognostic marker in cancer. Reduced cardiorespiratory fitness, measured objectively using cardiopulmonary exercise testing (CPET), is associated with higher perioperative risk, increased treatment-related complications, and poorer quality of life. Previous work from the study team and others has shown that chemotherapy and chemoradiotherapy for oesophageal and rectal cancer lead to significant declines in CPET-derived fitness, and that prescribed exercise prehabilitation can attenuate or reverse these declines and improve clinical outcomes.

Immune checkpoint inhibitors have become standard of care for a growing range of solid tumours in both adjuvant and metastatic settings. Immunotherapy is associated with distinct patterns of toxicity, including immune-related adverse events and cumulative treatment-related side effects that can impair day-to-day functioning, result in treatment delays, or lead to early discontinuation. However, the impact of immunotherapy on objectively measured physical fitness, and the extent to which baseline fitness and changes in fitness relate to toxicity, quality of life, and long-term outcomes, remains poorly defined.

Emerging evidence suggests complex interactions between physical fitness, immune function, and tumour biology. Exercise can influence systemic immunity and the tumour microenvironment, including increased infiltration of cytotoxic T cells and modulation of myeloid populations. These effects may help convert immunologically "cold" tumours with limited immune cell infiltration into "hot" tumours that are more responsive to immunotherapy. Understanding how baseline fitness and natural changes in fitness during immunotherapy relate to treatment tolerance and tumour-immune characteristics is therefore an important step towards rationally developing exercise-based interventions as potential adjuncts to immunotherapy.

This Phase II window observational study is a prospective, single-centre cohort study with an embedded mechanistic sub-study. It will enrol adults with histologically confirmed solid malignancies who are starting standard-of-care immune checkpoint inhibitor therapy at University Hospital Southampton NHS Foundation Trust. The trial adopts a tumour-agnostic approach, stratifying participants by treatment setting (adjuvant vs metastatic/palliative) and immunotherapy regimen (single-agent vs dual-agent checkpoint inhibition). This reflects real-world practice and allows evaluation of how treatment context and intensity influence changes in fitness and attrition.

For the observational cohort, participants will undergo baseline assessments within approximately two weeks prior to starting immunotherapy. These include CPET on a cycle ergometer to determine oxygen uptake at the anaerobic threshold (VO₂ at AT; primary outcome) and other CPET parameters, a panel of validated questionnaires assessing cancer-specific and generic quality of life, psychological distress, fatigue, social support and functional impact, grip strength, frailty assessment, targeted blood sampling (including nutritional markers, immune and metabolic biomarkers, and redox-related analytes), and review of standard-of-care imaging. Baseline medical history, comorbidities, and performance status will also be recorded.

During the first 12 weeks of immunotherapy, all anti-cancer treatment will be delivered according to usual clinical practice, independent of study participation. The research team will prospectively collect data on immunotherapy regimens (drug, dose, schedule), immune-related and treatment-related adverse events graded using CTCAE v5.0 and Society for Immunotherapy of Cancer (SITC) criteria, treatment delays, dose modifications, permanent or temporary discontinuations, and health-care utilisation such as unplanned admissions.

At approximately 12 weeks after immunotherapy initiation, participants will repeat the baseline battery of assessments: CPET, quality-of-life and psychosocial questionnaires, blood sampling, and documentation of treatment status. Radiological response will be evaluated using immune-adapted RECIST criteria on standard-of-care cross-sectional imaging where available. Participants will then enter long-term follow-up at approximately 6, 12, and 24 months from treatment start. Follow-up focuses on survival status, disease progression, ongoing treatment and toxicity, healthcare utilisation, repeated quality-of-life assessments, and selected clinical and nutritional measures. Questionnaires may be completed electronically, by telephone, or on paper, with a structured contact schedule to maximise response while respecting participant autonomy.

An optional mechanistic sub-study will invite up to 10 participants to undergo a research tumour biopsy at around 12 weeks, in addition to use of surplus baseline diagnostic biopsy material where consent permits. Research biopsies will be obtained via image-guided percutaneous procedures or endoscopy, depending on tumour location and standard diagnostic pathways. Recruitment to the mechanistic component will be stratified by tumour immunogenicity (for example, tumours with higher versus lower mutational burden and immune infiltration) to facilitate comparison across immunologically "hot" and "cold" tumours. Tumour tissue will undergo multiplex immunohistochemistry and complementary molecular profiling to characterise the tumour and immune microenvironment, including quantification of key immune cell subsets (such as CD8⁺ T cells, CD4⁺ subsets, regulatory T cells, and myeloid populations), checkpoint marker expression, and spatial organisation. Parallel blood samples will be used to explore systemic redox biology, metabolic flexibility, and immune signatures. All samples will be pseudonymised and stored in a Human Tissue Authority-licensed tissue bank according to predefined governance procedures for up to ten years, to enable further ethically approved analyses.

The observational component uses a precision-based sample size strategy. A total of 67 participants will be recruited across three strata, with 51 expected to contribute paired baseline and 12-week CPET data after accounting for differential attrition: adjuvant single-agent (20 recruited, 17 analysed), metastatic/palliative single-agent (23 recruited, 17 analysed), and metastatic/palliative dual-agent therapy (24 recruited, 17 analysed). This sample size allows estimation of mean change in VO₂ at AT with acceptable precision, with the overall 95% confidence interval spanning approximately ±0.55 standard deviations. Using planning values informed by prior exercise-oncology work (SD of change ≈1.8 mL/kg/min), 51 paired observations provide high power to detect a clinically important change of 1.5 mL/kg/min in VO₂ at AT, while recognising that the study is primarily exploratory and not powered for definitive hypothesis testing. The study will also estimate feasibility metrics such as recruitment, retention and completion of key assessments.

The primary analysis will describe changes in CPET-derived fitness between baseline and 12 weeks of immunotherapy, using paired tests for within-participant change and stratified analyses by treatment setting and regimen. Secondary and exploratory analyses will examine changes in other CPET parameters, the incidence and pattern of immunotherapy-related toxicity and treatment discontinuation during the first 12 weeks, trajectories of quality-of-life and psychosocial outcomes, and longer-term survival and disease control up to 24 months. Associations between baseline fitness and subsequent toxicity, treatment modification, quality of life, and survival will be explored using appropriate regression and time-to-event methods. Mechanistic analyses will integrate tumour, blood, and clinical data using largely non-parametric and multivariable approaches to generate biologically plausible effect size estimates and hypotheses for future studies; these analyses are explicitly exploratory.

Data will be collected in a secure, password-protected REDCap database with role-based access controls. CPET data will be processed according to standardised protocols, with key parameters independently reviewed by two exercise physiologists to support data quality. Routine data checks, range and consistency checks, and monitoring of recruitment and follow-up completeness will be undertaken by the trial team. Missing data will be described, and appropriate statistical methods for incomplete follow-up will be used where relevant; no complex imputation is planned for the primary outcome in this early-phase exploratory study.

The study was developed with input from a patient and public involvement and engagement (PPIE) group comprising individuals with lived experience of cancer. They contributed to decisions on study burden and acceptability, including the timing and mode of assessments, communication around optional biopsies, and support for travel costs. Their feedback informed participant materials and recruitment strategies, and ongoing involvement is planned during study delivery and dissemination.

Overall, this observational window study will characterise how immunotherapy affects objectively measured physical fitness and quality of life, clarify whether baseline fitness and early changes in fitness relate to toxicity and long-term outcomes, and provide mechanistic insight into links between fitness, immunotherapy, and the tumour microenvironment. These data are intended to define the natural history of fitness during immunotherapy, confirm that this represents a clinically meaningful problem, and provide the clinical and biological parameters needed to design a subsequent feasibility and effectiveness trial of structured exercise during immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed solid malignancy
* Receiving immune checkpoint inhibitors in one of the following settings:

  * Adjuvant: Single-agent anti-PD-1, anti-PD-L1, or anti-CTLA-4
  * Metastatic/Palliative: Single-agent or dual-agent anti-PD-1, anti-PD-L1, or anti-CTLA-4
* ECOG Performance Status 0-2
* Able to perform cardiopulmonary exercise testing
* Able to provide written informed consent
* Willing and able to comply with study procedures and follow-up schedule

Exclusion Criteria:

* Age <18 years
* Prior systemic anti-cancer immunotherapy for unresectable or metastatic disease, EXCEPT:
* Prior adjuvant or neoadjuvant immunotherapy if all treatment-related adverse events have returned to baseline or stabilized
* Prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy with at least 6 months since last dose and date of disease recurrence
* Absolute contraindications to cardiopulmonary exercise testing:
* Acute myocardial infarction within 6 weeks
* Unstable angina
* Uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise
* Active endocarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolism or pulmonary infarction
* Acute myocarditis or pericarditis
* Suspected or known dissecting aneurysm
* Acute systemic infection
* Inability to perform cardiopulmonary exercise testing (e.g., severe lower limb dysfunction, severe peripheral vascular disease)
* Inability to provide informed consent
* Currently enrolled in another interventional clinical trial that would confound study outcomes

ADDITIONAL EXCLUSION CRITERIA FOR RESEARCH BIOPSY SUB-STUDY:

* Severe cardiopulmonary disease precluding safe sedation (for endoscopic biopsies)
* Suspected bowel obstruction or perforation (for gastrointestinal biopsies)
* Uncorrectable severe coagulopathy (INR >1.5, platelet count <50,000/µL)
* Severe portal hypertension with high-risk varices (for upper endoscopy)
* Lesion inaccessible for safe biopsy as determined by a performing clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged ≥18 years with histologically confirmed solid malignancies receiving immune checkpoint inhibitors (anti-PD-1, anti-PD-L1, or anti-CTLA-4) at University Hospital Southampton. Recruitment includes patients treated in the adjuvant setting with single-agent therapy after definitive local treatment, and patients in the metastatic or palliative setting receiving single- or dual-agent immunotherapy for advanced disease. The study uses a tumour-agnostic approach and includes any solid tumour for which immunotherapy is indicated. Examples include gastrointestinal, thoracic, skin, genitourinary, gynaecological, head and neck, breast, and other solid cancers treated with checkpoint inhibitors. Participants must have ECOG Performance Status 0-2 and be able to safely undertake cardiopulmonary exercise testing.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oxygen Uptake at Anaerobic Threshold (VO₂ at AT) | Baseline and Week 12
  Change in oxygen uptake at the anaerobic threshold measured using cardiopulmonary exercise testing (CPET). VO₂ at AT will be reported in millilitres per kilogram per minute (mL·kg-¹·min-¹).

SECONDARY OUTCOMES:
Change in peak oxygen uptake (VO₂peak) | Baseline and Week 12
  Change in peak oxygen uptake measured during CPET. Unit: mL·kg-¹·min-¹
Change in peak power output | Baseline and 12 weeks
  Peak power output measured during CPET, reported in watts (W).
Change in ventilatory efficiency (VE/VCO₂ slope) | Baseline and week 12
  Ventilatory efficiency measured during CPET, reported as VE/VCO₂ slope (unitless ratio).
Cumulative Incidence of Immune-Related Adverse Events | Baseline (start of immunotherapy) through Month 24
  Cumulative incidence of immunotherapy-related toxicity graded using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and Society for Immunotherapy of Cancer (SITC) immune-related adverse event criteria. Captured through systematic review during treatment phase. reported as CTCAE grade and/or proportion of participants with ≥Grade 3 toxicity (%).
Treatment-Related Adverse Events Leading to Discontinuation | Baseline through Month 24
  Proportion of participants discontinuing immunotherapy due to treatment-related toxicity, reported as a percentage of participants (%).
Change in cancer-specific quality of life | Baseline, Week 12, Month 6, Month 12, and Month 24
  Cancer-specific quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) Global Health Status/QoL score. Unit of Measure: Score on a scale (0-100). Scale Details: 0 = worst quality of life, 100 = best quality of life. Higher scores indicate better quality of life.
Change in general health status | Baseline, Week 12, Month 6, Month 12, and Month 24
  General health status assessed using the EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) index score. Unit of Measure: Index score.
  Scale Details:
  Index values typically range from <0 (health states worse than death) to 1 (perfect health) Higher scores indicate better health status
Change in psychological distress | Baseline, Week 12, Month 6, Month 12, and Month 24
  Psychological distress assessed using the National Comprehensive Cancer Network (NCCN) Distress Thermometer. Unit of Measure: Score on a numeric rating scale (0-10)
  Scale Details:
  0 = no distress 10 = extreme distress Higher scores indicate worse distress
Change in anxiety and depression symptoms | Baseline, Week 12, Month 6, Month 12, and Month 24
  Anxiety and depression symptoms assessed using the Patient Health Questionnaire-4 (PHQ-4). Unit of Measure: Total score
  Scale Details:
  Range 0-12 Higher scores indicate greater anxiety and depressive symptoms
Change in fatigue severity | Baseline, Week 12, Month 6, Month 12, and Month 24
  Fatigue severity assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form: reported as T-score (mean 50), higher scores indicate worse fatigue.
Change in perceived social support | Baseline, Week 12, Month 6, Month 12, and Month 24
  Modified Medical Outcomes Study Social Support Survey (mMOS-SSS); score range 0-100, higher scores indicate greater support.
Change in functional impairment | Baseline, Week 12, Month 6, Month 12, Month 24
  Work and Social Adjustment Scale (WSAS); total score range 0-40, higher scores indicate worse impairment.
Change in functional capacity | Baseline, Week 12, Month 6, Month 12, Month 24
  Duke Activity Status Index (DASI); score range 0-58.2, higher scores indicate better functional capacity
Change in frailty status | Baseline, Week 12, Month 6, Month 12, Month 24
  Edmonton Frail Scale (EFS); total score range 0-17, higher scores indicate worse frailty.
Recruitment feasibility | During recruitment period - 12 months
  Proportion of eligible participants who consent to the observational study, calculated as number consented divided by number screened, reported as percentage (%).
Adherence to research assessments | Baseline and Week 12
  Proportion of participants completing each scheduled research assessment (e.g. CPET, questionnaires), reported as percentage (%).
Feasibility of Optional Research Biopsy | Week 12
  Proportion of participants who consent to and complete the optional Week-12 research biopsy, reported as a percentage (%).
Biopsy-related complications | Week 12
  Proportion of participants experiencing biopsy-related complications following the optional Week-12 research biopsy, reported as a percentage (%).

OTHER OUTCOMES:
Overall survival | Baseline (start of immunotherapy) through 24 months of follow-up
  Time from initiation of immunotherapy to death from any cause, assessed using routine clinical follow-up and medical records.
Disease-free survival | Baseline (start of immunotherapy) through 24 months of follow-up
  Time from initiation of immunotherapy to first documented disease recurrence, progression, or death from any cause, assessed using routine clinical follow-up and imaging. Unit of Measure: Time (months)
Event-free survival | Baseline (start of immunotherapy) through 24 months of follow-up
  Time from initiation of immunotherapy to disease progression, treatment discontinuation due to disease progression or treatment-related toxicity, or death from any cause, whichever occurs first, assessed using routine clinical follow-up and imaging. Unit of Measure: Time (months)
Disease progression status | At 6, 12, and 24 months following initiation of immunotherapy
  Presence or absence of disease progression assessed using routine clinical imaging and clinical follow-up according to standard-of-care criteria. Unit of Measure: Categorical (progression / no progression)
Change in nutritional status | Baseline to 12 months
  Nutritional status assessed using the Patient-Generated Subjective Global Assessment (PG-SGA); total score, higher scores indicate worse nutritional status.
Health economic outcomes | Baseline through Month 24
  Healthcare utilisation (e.g. admissions, visits) reported as counts and/or costs (GBP).
Radiologic Response to Immunotherapy | Baseline and Week 12
  Radiological tumour response assessed by study radiologist using immune RECIST (iRECIST) criteria: iCR (complete response), iPR (partial response), iSD (stable disease), iUPD (unconfirmed progressive disease), iCPD (confirmed progressive disease), or NE (not evaluable). Applies to metastatic setting only.
Change in tumour immune marker expression (Mechanistic Sub-Study) | Baseline diagnostic biopsy and optional week-12 research biopsy
  Tumour immune marker expression quantified using immunohistochemistry on baseline diagnostic biopsy and optional Week-12 research biopsy tissue; reported as percentage of positively stained cells (%).
Change in tumour gene expression signatures | Baseline diagnostic biopsy and optional Week-12 biopsy
  Tumour molecular signatures measured using bulk RNA sequencing; results summarised as unitless pathway or gene-signature scores derived from normalised expression data.
Association between fitness and tumour/biological markers | Baseline and Week 12
  Association between physical fitness, measured by oxygen uptake at anaerobic threshold (VO₂ at AT) from cardiopulmonary exercise testing (CPET, mL·kg-¹·min-¹), and tumour or blood-based biological markers previously defined in this study.
  Associations will be reported using correlation or regression effect estimates between VO₂ at AT and tumour immune marker expression (immunohistochemistry, % positive cells), tumour gene expression signatures (bulk RNA sequencing, unitless signature scores), and a composite redox/metabolic biomarker index (unitless composite score).
Change in composite redox and metabolic biomarker index | Change in a pre-specified composite index reflecting systemic redox balance and metabolic flexibility, derived from standardised (z-score normalised) circulating blood-based biomarkers; unitless composite score.
  Change in composite redox a

CONTACTS AND LOCATIONS:
Overall Officials: Kashuf Khan, MBBS, MRCS, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie published results will be made available after deidentification, including data dictionary. Access will be granted to researchers whose proposed use has been approved by an independent review committee for methodologically sound proposals achieving aims in the approved proposal.
  Proposals should be directed to m.west@soton.ac.uk and will require a data access agreement. Data will be available beginning 12 months and ending 5 years following article publication.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Kurz E, Hirsch CA, Dalton T, Shadaloey SA, Khodadadi-Jamayran A, Miller G, Pareek S, Rajaei H, Mohindroo C, Baydogan S, Ngo-Huang A, Parker N, Katz MHG, Petzel M, Vucic E, McAllister F, Schadler K, Winograd R, Bar-Sagi D. Exercise-induced engagement of the IL-15/IL-15Ralpha axis promotes anti-tumor immunity in pancreatic cancer. Cancer Cell. 2022 Jul 11;40(7):720-737.e5. doi: 10.1016/j.ccell.2022.05.006. Epub 2022 Jun 2. PMID 35660135
- [Background] Wennerberg E, Lhuillier C, Rybstein MD, Dannenberg K, Rudqvist NP, Koelwyn GJ, Jones LW, Demaria S. Exercise reduces immune suppression and breast cancer progression in a preclinical model. Oncotarget. 2020 Jan 28;11(4):452-461. doi: 10.18632/oncotarget.27464. eCollection 2020 Jan 28. PMID 32064049
- [Background] Maleki Vareki S. High and low mutational burden tumors versus immunologically hot and cold tumors and response to immune checkpoint inhibitors. J Immunother Cancer. 2018 Dec 27;6(1):157. doi: 10.1186/s40425-018-0479-7. PMID 30587233
- [Background] Kong X, Chen L, Su Z, Sullivan RJ, Blum SM, Qi Z, Liu Y, Huo Y, Fang Y, Zhang L, Gao J, Wang J. Toxicities associated with immune checkpoint inhibitors: a systematic study. Int J Surg. 2023 Jun 1;109(6):1753-1768. doi: 10.1097/JS9.0000000000000368. PMID 37132038
- [Background] Kennedy LB, Salama AKS. A review of cancer immunotherapy toxicity. CA Cancer J Clin. 2020 Mar;70(2):86-104. doi: 10.3322/caac.21596. Epub 2020 Jan 16. PMID 31944278
- [Background] McIsaac DI, Gill M, Boland L, Hutton B, Branje K, Shaw J, Grudzinski AL, Barone N, Gillis C; Prehabilitation Knowledge Network. Prehabilitation in adult patients undergoing surgery: an umbrella review of systematic reviews. Br J Anaesth. 2022 Feb;128(2):244-257. doi: 10.1016/j.bja.2021.11.014. Epub 2021 Dec 16. PMID 34922735
- [Background] West MA, Baker WC, Rahman S, Munro A, Jack S, Grocott MP, Underwood TJ, Levett DZ; Fit-4-Surgery Consortium. Cardiopulmonary exercise testing has greater prognostic value than sarcopenia in oesophago-gastric cancer patients undergoing neoadjuvant therapy and surgical resection. J Surg Oncol. 2021 Dec;124(8):1306-1316. doi: 10.1002/jso.26652. Epub 2021 Aug 31. PMID 34463378
- [Background] Loughney LA, West MA, Kemp GJ, Grocott MP, Jack S. Exercise interventions for people undergoing multimodal cancer treatment that includes surgery. Cochrane Database Syst Rev. 2018 Dec 11;12(12):CD012280. doi: 10.1002/14651858.CD012280.pub2. PMID 30536366
- [Background] West MA, Loughney L, Barben CP, Sripadam R, Kemp GJ, Grocott MP, Jack S. The effects of neoadjuvant chemoradiotherapy on physical fitness and morbidity in rectal cancer surgery patients. Eur J Surg Oncol. 2014 Nov;40(11):1421-8. doi: 10.1016/j.ejso.2014.03.021. Epub 2014 Apr 12. PMID 24784775
- [Background] Loughney L, West MA, Moyses H, Bates A, Kemp GJ, Hawkins L, Varkonyi-Sepp J, Burke S, Barben CP, Calverley PM, Cox T, Palmer DH, Mythen MG, Grocott MPW, Jack S; Fit4Surgery group. The effects of neoadjuvant chemoradiotherapy and an in-hospital exercise training programme on physical fitness and quality of life in locally advanced rectal cancer patients: a randomised controlled trial (The EMPOWER Trial). Perioper Med (Lond). 2021 Jun 22;10(1):23. doi: 10.1186/s13741-021-00190-8. PMID 34154675
- [Background] Steffens D, Ismail H, Denehy L, Beckenkamp PR, Solomon M, Koh C, Bartyn J, Pillinger N. Preoperative Cardiopulmonary Exercise Test Associated with Postoperative Outcomes in Patients Undergoing Cancer Surgery: A Systematic Review and Meta-Analyses. Ann Surg Oncol. 2021 Nov;28(12):7120-7146. doi: 10.1245/s10434-021-10251-3. Epub 2021 Jun 8. PMID 34101066
- [Background] Hapuarachi B, Danson S, Wadsley J, Muthana M. Exercise to transform tumours from cold to hot and improve immunotherapy responsiveness. Front Immunol. 2023 Dec 12;14:1335256. doi: 10.3389/fimmu.2023.1335256. eCollection 2023. PMID 38149260